CLINICAL TRIAL: NCT02077374
Title: A Placebo-Controlled, Multicenter, Double-Blind, Randomized Trial of IDN-6556 in Subjects With Non-Alcoholic Fatty Liver Disease and Raised Transaminases
Brief Title: A Study of IDN-6556 in Subjects With NAFLD and Raised Transaminases
Acronym: NAFLD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Conatus Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IDN-6556-06
Record Dates: First submitted 2014-02-28; First posted 2014-03-04 (Estimated); Results first posted 2016-07-21 (Estimated); Last update posted 2016-08-30 (Estimated); Status verified 2016-07

CONDITIONS: Nonalcoholic Steatohepatitis; Non-alcoholic Fatty Liver Disease
Keywords: NAFLD; NASH
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — 3-(2-(2-tert-butylphenylaminooxalyl)aminopropionylamino)-4-oxo-5-(2,3,5,6-tetrafluorophenoxy)pentanoic acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IDN-6556 (Experimental): IDN-6556 capsules, 25 mg BID
  Interventions: Drug: IDN-6556
- Placebo (Placebo Comparator): Placebo BID
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: IDN-6556 — 25 mg BID for 28 days
  Other Names: emricasan; PF-03491390
  Arms: IDN-6556
Other: Placebo — Placebo BID for 28 Days
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the safety and efficacy of IDN-6556 compared to placebo in patients with diagnosed fat deposits in their liver (not caused by alcohol) and with abnormal liver tests

DETAILED DESCRIPTION:
This is a double-blind, randomized study to evaluate the effects of IDN-6556 on serum transaminases and pharmacodynamics of IDN-6556 in subjects with non-alcoholic fatty liver disease with elevated alanine aminotransferase.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects of minimum adult legal age (according to local laws for signing the informed consent document), able to provide written informed consent, and understand and comply with the requirements of the study
* Diagnosis of non-alcoholic fatty liver disease (NAFLD) as evidenced by imaging or other diagnostic assessments
* Alanine aminotransferase (ALT) levels ≥1.5 x ULN on at least two occasions, seven or more days apart, during the Screening period
* alpha-fetoprotein (AFP) ≤ 100 ng/mL
* Hemoglobin ≥10 g/dL, a platelet count ≥ 100 x 10^9/L, and a white blood cell count ≥ 3.0 x 10^9/L
* If on metformin, sulfonylureas, statins, or fibrates, subjects must be on a stable dose of these drugs for at least three months prior to Screening and during the study

Exclusion Criteria:

* Known infection with HIV, HCV, or HBV
* Decompensated or severe liver disease as evidenced by one or more of the following:

  1. Confirmed cirrhosis or suspicion of cirrhosis
  2. Esophageal varices
  3. Ascites
  4. Suspicion of portal hypertension
  5. Hospitalization for liver disease within 60 days of screening
  6. Bilirubin >2 x ULN, or ALT or AST > 10 x ULN
* Inflammatory bowel disease
* Diagnosed or suspected systemic lupus erythematosus (SLE) and/or rheumatoid arthritis (RA)
* Hepatocellular carcinoma (HCC) at entry into the study
* History of or active non-liver malignancies other than curatively treated skin cancer (basal cell or squamous cell carcinomas)
* Significant systemic or major illness other than liver disease, including coronary artery disease, cerebrovascular disease, pulmonary disease, renal insufficiency, and/or serious psychiatric disease, that, in the opinion of the Investigator would preclude the subject from participating in and completing the study
* History or presence of alcohol abuse, defined as consumption of more than 210 mL of alcohol per week (the equivalent of 14 4-ounce glasses of wine or 14 12-ounce cans/bottles of beer or wine coolers), or other substance abuse within the prior two years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2014-03; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean L. Chan, MD, Study Director — Conatus Pharmaceuticals Inc.
Locations (7):
- United States (7):
  - University of Miami, Miami, Florida
  - Indiana University, Indianapolis, Indiana
  - Henry Ford Hospital, Detroit, Michigan
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Kansas City Research Institute, Kansas City, Missouri
  - Mary Immaculate Hospital, Newport News, Virginia
  - Bon Secours St. Mary's Hospital, Richmond, Virginia

REFERENCES:
- [Derived] Shiffman M, Freilich B, Vuppalanchi R, Watt K, Chan JL, Spada A, Hagerty DT, Schiff E. Randomised clinical trial: emricasan versus placebo significantly decreases ALT and caspase 3/7 activation in subjects with non-alcoholic fatty liver disease. Aliment Pharmacol Ther. 2019 Jan;49(1):64-73. doi: 10.1111/apt.15030. Epub 2018 Nov 14. PMID 30430605

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In total, 71 subjects were screened at 7 sites, and 38 subjects were randomized and treated to a BID treatment with either placebo or IDN-6556 25 mg with 19 subjects in each arm.
Pre-assignment Details: 38 subjects were randomized and treated (19 each arm). 2 subjects on placebo discontinued before Day 28 and 1 discontinued after Day 28, but returned for their Day 56 visit, so 17 subjects completed the study. However, all 38 were included in the analyses using the last results provided for the 2 subjects at early termination.
Groups:
- IDN-6556: IDN-6556 capsules, 25 mg
  IDN-6556: 25 mg BID for 28 days
- Placebo: Placebo
  Matching Placebo BID for 28 days
Period: Overall Study
Arm/Group | IDN-6556 | Placebo
Started | 19 | 19
Completed | 19 | 17
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IDN-6556 | Placebo | Total
Number analyzed (Participants) | 19 | 19 | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 16 | 33
  >=65 years | 2 | 3 | 5
Age, Continuous [Median (Full Range); unit: years] | 46 [23 to 76] | 55 [34 to 70] | 52 [23 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 14
  Male | 12 | 12 | 24
Region of Enrollment [Number; unit: participants]
  United States | 19 | 19 | 38

OUTCOME MEASURES:

1. Primary Outcome: Change in Alanine Aminotransferase (ALT)
Description: Mean change in alanine aminotransferase (ALT) from Baseline to Day 28/ET between IDN-6556 vs Placebo
Time Frame: Day 28/ET
Population: The full analysis set (FAS) included all subjects who were randomized and received at least one dose of study drug. For the FAS, subjects were assigned to the treatment group based on the randomization schedule, regardless of the treatment they actually received. All efficacy analyses were conducted on the FAS.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | IDN-6556 | Placebo
Number analyzed (Participants) | 19 | 19
U/L | -37.8 (42.7) | -14.9 (22.5)
Statistical Analysis 1: Comparison: IDN-6556 vs Placebo; Statistical Analysis for the difference in mean change in alanine aminotransferase (ALT) from Baseline to Day28/ET between IDN-6556 and placebo; Test type: Superiority or Other; p = 0.0195, Wilcoxon (Mann-Whitney); Mean Difference (Net) = -17, 95% CI 2-sided [-30.7 to -2.5] — Based on Hodges-Lehmann estimator

2. Primary Outcome: Relative Percent Change in Alanine Aminotransferase (ALT)
Description: Back transformation from log-transformed analysis results to original scale in alanine aminotransferase (ALT) from Baseline to Day 28/ET between IDN-6556 vs Placebo
Time Frame: Baseline to Day 28/ET
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Relative percent change
Groups:
- IDN-6556: IDN-6556 capsules, 25 mg
  IDN-6556: 25 mg Twice daily for 28 days
- Placebo: Placebo
  Placebo: Placebo Twice daily for 28 Days
Arm/Group | IDN-6556 | Placebo
Number analyzed (Participants) | 19 | 19
Relative percent change | -39.2 (26.2) | -13.9 (21.8)

3. Secondary Outcome: Change in Aspartate Aminotransferase (AST)
Description: Difference in the change in aspartate aminotransferase (AST) from Baseline to Day 28/ET in units per liter (U/L) between IDN-6556 and placebo.
Time Frame: Day 28/ET
Population: as for outcome 1
Measure: Median (Full Range); unit: U/L
Arm/Group | IDN-6556 | Placebo
Number analyzed (Participants) | 19 | 19
U/L | -6.7 [-63.1 to 20.0] | -5.2 [-41.9 to 27.9]
Statistical Analysis 1: Comparison: IDN-6556 vs Placebo; Statistical Analysis for the difference in change in aspartate aminotransferase (AST) from baseline to Day 28/ET between IDN-6556 and placebo; Test type: Superiority or Other; p = 0.8724, Wilcoxon (Mann-Whitney); Median Difference (Net) = -0.8, 95% CI 2-sided [-14.5 to 11.2] — Based on Hodges-Lehmann estimator

4. Secondary Outcome: Levels of cCK18/M30
Description: Difference in the change in Caspase-cleaved cytokeratin serum levels (cCK18/M30) in units per liter (U/L) from baseline to Day 28/ET between IDN-6556 and placebo
Time Frame: Day 28/ET
Population: as for outcome 1
Measure: Median (Full Range); unit: U/L
Arm/Group | IDN-6556 | Placebo
Number analyzed (Participants) | 19 | 19
U/L | -183.0 [-640 to 190] | 14.0 [-2056 to 571]
Statistical Analysis 1: Comparison: IDN-6556 vs Placebo; Statistical Analysis for the difference in change for cCK18/M30 from Baseline to Day 28/ET between IDN-6556 and Placebo; Test type: Superiority or Other; p = 0.1149, Wilcoxon (Mann-Whitney); Median Difference (Net) = -145, 95% CI 2-sided [-336 to 55] — Based on Hodges-Lehmann estimator

5. Secondary Outcome: Levels of Caspase 3/7 RLU
Description: Difference in the change of caspase 3/7 (Relative Light Units) from baseline to Day 28/ET between IDN-6556 and Placebo
Time Frame: Day 28/ET
Population: as for outcome 1
Measure: Median (Full Range); unit: RLU
Arm/Group | IDN-6556 | Placebo
Number analyzed (Participants) | 19 | 19
RLU | -287.0 [-2194 to 417] | 68.0 [-1779 to 1229]
Statistical Analysis 1: Comparison: IDN-6556 vs Placebo; Statistical Analysis for the difference in change for caspase 3/7 from Baseline to Day 28/ET between IDN-6556 and Placebo; Test type: Superiority or Other; p = 0.1365, Wilcoxon (Mann-Whitney); Median Difference (Net) = -250, 95% CI 2-sided [-590 to 63] — Based on Hodges-Lehmann estimator

6. Secondary Outcome: Levels of flCK18/M65
Description: Difference in the change in full-length cytokeratin 18 (flCK18/M65) in units per liter (U/L) from Baseline to Day 28/ET between IDN-6556 and placebo
Time Frame: Day 28/ET
Population: as for outcome 1
Measure: Median (Full Range); unit: U/L
Groups:
- Placebo: Placebo
  Placebo: Placebo BID for 28 Days
Arm/Group | IDN-6556 | Placebo
Number analyzed (Participants) | 19 | 19
U/L | -296.0 [-1216 to 225] | 4.0 [-2364 to 724]
Statistical Analysis 1: Comparison: IDN-6556 vs Placebo; Statistical Analysis of the difference in the change in full-length cytokeratine 18 (flCK18/M65) from Baseline to Day 28/ET between IDN-6556 and placebo; Test type: Superiority or Other; p = 0.0471, Wilcoxon (Mann-Whitney); Median Difference (Net) = -327, 95% CI 2-sided [-628 to -7] — Based on Hodges-Lehmann estimator

ADVERSE EVENTS:
Time Frame: Adverse events data were collected up to Day 56.
Arm/Group | IDN-6556 | Placebo
Serious Adverse Events (participants affected / at risk) | 1/19 | 1/19
Other Adverse Events (participants affected / at risk) | 10/19 | 8/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IDN-6556 (N=19) | Placebo (N=19)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cellulitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IDN-6556 (N=19) | Placebo (N=19)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Frequent bowel movements (Gastrointestinal disorders) | 2 (2) | 0 (0)
Chest pain (General disorders) | 2 (2) | 0 (0)
Injection site erythema (General disorders) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (2)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Monoclonal B-cell lymphocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 1 (1)
Injection site swelling (General disorders) | 0 (0) | 1 (1)
Local Swelling (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less